CLINICAL TRIAL: NCT03477500
Title: Randomized Autologous heMatopoietic Stem Cell Transplantation Versus Alemtuzumab, Cladribine or Ocrelizumab for Patients With Relapsing Remitting Multiple Sclerosis (RAM-MS)
Brief Title: Randomized Autologous heMatopoietic Stem Cell Transplantation Versus Alemtuzumab, Cladribine or Ocrelizumab for RRMS (RAM-MS)
Acronym: RAM-MS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-001362-25
Record Dates: First submitted 2018-02-13; First posted 2018-03-26 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis,; HSCT; alemtuzumab; RCT
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cyclophosphamide; Alemtuzumab; Cladribine; ocrelizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HSCT (Cyclophosphamide and ATG) (Experimental): Day 1: Cyclophosphamide 2.0 g/m2 body surface area Days 5-10: Granulocyte colony stimulating factor (filgrastim) 5 mcg/kg body weight/day sc.
  Day 11 and until apheresis is discontinued: Granulocyte colony stimulating factor (filgrastim) 5 mcg/kg body weight x 2 sc/day.
  HSCT days -5 to -2: Cyclophosphamide 50 mg/kg/day. HSCT days -5 to -1: Anti-thymocyte globulin (ATG-rabbit, Thymoglobuline®) 0.5 mg/kg body weight iv on day -5, 1.0 mg ATG-rabbit/kg will be given iv on day -4, and 1.5 mg ATG-rabbit /kg will be given iv on days -3,-2 and -1 over 10 hours.
  HSCT day 0: Reinfusion of a minimum of 3,0 x 106 CD 34+ cells/kg body weight.
  Interventions: Drug: Cyclophosphamide and ATG
- Alemtuzumab, Cladribine or Ocrelizumab (Active Comparator): Alemtuzumab, Cladribine or Ocrelizumab administered after the label of the study drug.
  Interventions: Drug: Alemtuzumab; Drug: Cladribine Pill; Drug: Ocrelizumab

INTERVENTIONS:
Drug: Cyclophosphamide and ATG — Hematopoetic stem cell transplantation
  Other Names: Sendoxan
  Arms: HSCT (Cyclophosphamide and ATG)
Drug: Alemtuzumab — Alemtuzumab (Lemtrada)
  Other Names: Lemtrada
  Arms: Alemtuzumab, Cladribine or Ocrelizumab
Drug: Cladribine Pill — Cladribine (Mavenclad)
  Other Names: Mavenclad
  Arms: Alemtuzumab, Cladribine or Ocrelizumab
Drug: Ocrelizumab — Ocrelizumab (Ocrevus)
  Other Names: Ocrevus
  Arms: Alemtuzumab, Cladribine or Ocrelizumab

SUMMARY:
This study is a randomized multicentre, multinational, treatment interventional study of RRMS patients with breakthrough inflammatory disease activity in spite of ongoing standard immunomodulatory medication. The study has two treatment arms; arm A: HSCT (hematopoietic stem cell transplantation) and arm B: alemtuzumab, cladribine or ocrelizumab. A pre-planned 3-year follow-up extension period will be performed depending on future funding.

The aim of the study is to assess the effectiveness and side effects of a new treatment intervention in RRMS; HSCT, and, thereby, the value of HSCT in clinical practice. Data from recently published patient series indicate that HSCT may have a significantly higher treatment effect than currently registered RRMS immunomodulatory treatments. This study will determine the relative role of HSCT versus alemtuzumab, cladribine or ocrelizumab.

DETAILED DESCRIPTION:
This is a randomized study of autologous HSCT using a low intensity, non-ablative conditioning regimen with cyclophosphamide and ATG versus treatment with the currently presumed best available immunomodulatory medication (alemtuzumab, cladribine or ocrelizumab) in RRMS patients with significant inflammatory disease activity in spite of ongoing immunomodulatory MS treatment.

Significant disease activity is defined as having one or more clinically reported multiple sclerosis (MS) relapse(s), AND 1 or more T1 Gd-enhanced lesion(s), OR three or more new or enlarging T2 lesions on magnetic resonance imaging (MRI) over the last year while being treated on immunomodulatory medication by standard national guidelines. The relapse(s) must have occurred 3 or more months after the onset of an immunomodulatory treatment, as immunomodulatory treatment in MS may reach full effect after 3 months or more.

Both the knowledge of the treatment effect of registered immunomodulatory therapies for RRMS, and the number of treatments approved for RRMS by the European Medicines Agency (EMA) are rapidly increasing. During the study period, there may thus appear new supplementing information on other MS immunomodulatory treatments that favour the use of a new comparator (replacing or supplementing the comparators). This will be evaluated by the PMC if applicable during the study period and the planned extension period.

If the treatment efficacy obtained by HSCT is better than the currently most efficacious standard, immunomodulatory treatment in randomized treatment trials, HSCT will likely be approved as a part of the standard treatment recommendations for a significant proportion of RRMS patients. A randomized study regarding with statistical power to evaluate the clinical outcome of autologous HSCT compared to a standard immunomodulatory treatment in MS has not yet been published. Except for Sweden, HSCT is currently not registered as a part of standard MS treatment in the public health services of Europe. The HSCT regimen for the study will be identical to the regimen used in similar patient populations in Sweden, Norway and Denmark.

Alemtuzumab, cladribine or ocrelizumab have been chosen as the primary comparators, because they are the immunomodulatory medication currently authorised by the EMA for treatment of RRMS with the most favourable therapeutic effects. In a meta-analysis of immunomodulatory treatment effects in RRMS, thse medications had the most eminent reduction of annualized relapse rate and 3 month confirmed disability progression.

In this study, a health economic evaluation will be included. Accordingly, the proposed study should provide a robust basis for future official decisions regarding the role of HSCT in RRMS treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between ≥18 to ≤50, both genders
2. Women of childbearing potential* (WOCBP) and men in a sexual relation with WOCBP must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.
3. Diagnosis of RRMS using revised McDonald criteria of clinically definite MS1
4. An EDSS score of 0 to 5.5
5. Significant inflammatory disease activity in the last year despite treatment with standard disease modifying therapy (interferon beta, glatiramer acetate, dimethyl fumarate, teriflunomide, fingolimod, natalizumab)

   a. Significant inflammatory disease activity is defined by: i. One or more clinically reported multiple sclerosis (MS) relapse(s), ii. AND 1 or more T1 Gd-enhanced lesion(s), iii. OR three or more new or enlarging T2 lesions on magnetic resonance imaging (MRI) The relapse(s) must have been treated with iv or oral high dose corticosteroids prescribed by a neurologist, and must have occurred 3 or more months after the onset of an immunomodulatory treatment, as MS immunomodulatory treatment may reach full effect after 3 months or more2.
6. The patient is a RRMS-patient referred from neurological departments in Norway, Denmark, Sweden or possibly other European countries to an assigned study site.
7. Signed informed consent and expected patient cooperation regarding the treatment schemes and procedures planned in the treatment and follow-up periods must be obtained and documented according to ICH GCP and national/local regulations.

Exclusion Criteria:

1. Known hypersensitivity or other known serious side effects for any of the study medications, including co-medications such as high-dose glucocorticosteroids
2. Any illness or prior treatment that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemotherapy or high-dose glucocorticosteroids
3. Any ongoing infection, including Tbc, CMV, EBV, HSV, VZV, hepatitis virus, toxoplasmosis, HIV or syphilis infections, as well as heaptitis B surface antigen positivity and/or hepatitis C PCR positivity verified at Visit 1
4. Patients without a history of chickenpox or without vaccination against varicella zoster virus (VZV), unless tested for antibodies to VZV. VZV negative patients can only be included if they receive vaccination against VZV at least 6 weeks prior to inclusion.
5. Current or previous treatments with long-term effects that may influence the treatment effects or potential toxicities/side effects of the treatment arms. This includes, but is not restricted to previous treatment with rituximab, mitoxantrone, alemtuzumab, cladribin and ocrelizumab
6. Immunocompromised patients, or patients currently reveiving immunosuppressive or myelosuppressive therapy
7. Treatment with glucocorticoids or ACTH within one month prior to start of study treatment
8. Having experienced an MS relapse within one month prior to study inclusion
9. Prior or current major depression
10. Prior or current psychiatric illness, mental deficiency or cognitive dysfunction influencing the patient ability to make an informed consent or comply with the treatment and follow-up phases of this protocol.
11. Prior or current alcohol or drug dependencies
12. Cardiac insufficiency, cardiomyopathy, significant cardiac dysrhytmia, unstable or advanced ischemic heart disease (NYHA III or IV)
13. Significant hypertension: BP > 180/110
14. Active malignancy, or prior history of malignancy except localized basal cell, squamous skin cancer or carcinoma in situ of the cervix.
15. Known untreated or unregulated thyroid disease
16. Failure to willingly accept or comprehend risk of irreversible sterility as a side effect of therapy
17. WBC < 1,5 x 109/L if not caused by a reversible effect of documented ongoing medication. If WBC < 1,5 x 109/L is caused by a reversible effect of documented ongoing medication the WBC count must be > 1,5 x 109/L before start of study treatment.
18. Platelet (thrombocyte) count < 100 x 109/L
19. ALAT and/or ASAT more than 2 times the upper normal reference limit (UNL)
20. Serum creatinine > 200 µmol/L
21. Serum bilirubin > ULN
22. Moderate or severely impaired kidney function (creatinine-clearance below 60 ml/min)
23. Presence of metallic objects implanted in the body that would preclude the ability of the patient to safely have MRI exams
24. Diagnosis of primary progressive MS
25. Diagnosis of secondary progressive MS
26. Treatment with natalizumab and fingolimod within the last 2 months, and treatment with dimetylfumurat within the last month (washout must be performed as specified in section 5.1) prior to start of study medication.
27. Use of teriflunomide (Aubagio®) within the previous 2 years unless cleared from the body (plasma concentration < 0.02 mcg/ml following elimination from the body with cholestyramine or activated powdered charcoal) as specified in section 5.1 prior to start of study medication.
28. Any hereditary neurological disease such as Charcot-Marie-Tooth disease or Spinocerebellar ataxia
29. Any disease that can influence the patient safety and compliance, or the evaluation of disability
30. History of hypersensitivity reaction to rabbit
31. Women who are pregnant, breast-feeding, or who plan to become pregnant within the timeframe of this study
32. Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational treatment(s). Patients participating in a purely observational trial will not be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-21 (Actual); Primary Completion 2026-11-21 (Estimated); Study Completion 2028-03-21 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with no evidence of disease activity (NEDA, as defined per protocol). | 2 year (96 week) period with a 5 year (240 week) planned extension
  A protocol-defined disease activity event is the occurrence of at least one of the following:
  * A new T1 Gd-enhanced lesion on MRI of the brain and spinal cord
  * A new T2 hyperintense lesion on MRI of brain and spinal cord
  * A protocol-defined MS relapse (see below)
  * 24 week confirmed disability progression based on increases in Expanded Disability Status Scale (EDSS)

SECONDARY OUTCOMES:
NEDA-4 | 2 year (96 week) period
  Proportion of patients with no evidence of disease activity, including atrophy (NEDA 4), as per protocol defined disease activity events (as defined in section 2.2) plus atrophy (measured yearly atrophy above threshold of 0, 4 %)
Pre-planned study extension: | 5 year (240 week) period.
  Proportion of patients who have NEDA 4
Time to first protocol-defined disease activity event | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Time to first sign of new disease activity, as measured as new relapses, EDSS-progression, MRI-activity or brain atrophy
Change in Expanded Disability Status scale (EDSS) from baseline (Visit 4.1) to Weeks 96 and 240 | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses the 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), where higher scores indicate worse neurological function. Change was calculated by subtracting retreatment baseline (annual visit prior to the retreatment start date) value from EDSS scores at specified time points.
The proportion of patients who, at Week 96, have protocol-defined Confirmed Disability Improvement (CDI) , confirmed stable EDSS or Confirmed Disability Progression (CDP) compared to baseline | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Disability progression, as measured with EDSS. EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses the 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), where higher scores indicate worse neurological function. Change was calculated by subtracting retreatment baseline (annual visit prior to the retreatment start date) value from EDSS scores at specified time points.
Annualized rate of protocol-defined relapses during 96 weeks | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  ARR
Time to onset of first protocol-defined relapse | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Time to first relapse
Change in MRI T2-weighted hyperintense lesion volume from baseline to weeks 96 (and 240) | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Change in T2-weighted hyperintense lesion volume
Change in MRI T1-weighted hypointense lesion volume from baseline to weeks 96 (and 240) | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Change in MRI T1-weighted hypointense lesion volume
Change in brain volume from baseline to week 96 (and week 240) | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Change in brain volume
Time to detection of a new MRI T2 lesion | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Time to New MRI T2-lesion
Total number of MRI T1-weighted Gd-enhanced lesions | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Number of Gd-lesions
Proportion of patients free from T1 Gd-enhancing lesions | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Proportion of patients free from T1 Gd-enhancing lesions
Change in Nine-hole-peg test (9-HPT) score from baseline to week 96 (and 240) | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  The 9HPT is a brief, standardized, quantitative test of upper extremity function. The participant picks up 9 pegs puts them in a block containing nine empty holes, and, once they are in the holes, removes them again as quickly as possible one at a time. The total time to complete the task is recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand. The two trials for each hand are averaged
Change in Timed 25 Foot Walk (T25FW) score from baseline to week 48, 96 (and 240) | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  The T25FW is a quantitative mobility and leg function performance test based on a timed walk over 25 feet. The participant is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the participant has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. The score for the T25FW is the average of the 2 completed trials. The 95% CI of the percentage is based on normal approximation.
Change in The Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) score from baseline to week 96 (and 240) | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  BICAMS is a composite cognitive assessment tool comprising of the three components : Symbol Digit Modalities Test (SDMT) , California Verbal Learning Test-II (CVLT-II) and Brief visuospatial memory test- Revised (BVMT-R)

OTHER OUTCOMES:
Difference in patient reported quality of life based on the EuroQoL Health Related Quality of Life - 5 Dimensions - 5 Levels (EQ-5D 5L) scores | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  EQ-5D 5L is a 5 item questionnaire (assessing - mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and visual analogue scale (VAS) enables calculation of quality adjusted life years (QALY) to enable health economic analyses to be performed. Each dimension assessed has 5 response scales to select from: no problems, slight problems, moderate problems, severe problems, and extreme problems
Overall survival rate | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Survival
Rate and nature of adverse events | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Rate and nature of adverse events
Fatigue Severity Scale (FSS) | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  The FSS questionnaire contains nine statements that rate the severity of fatigue symptoms. A low value (e.g., 1); indicates strong disagreement with the statement, whereas a high value (e.g., 7); indicates strong agreement. A total score of 36 or more suggests presence of fatigue.
Change in Multiple Sclerosis Impact Scale (MSIS) - 29 | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Multiple Sclerosis Impact Scale-29 (MSIS-29) is a validated MS specific questionnaire consisting of 29 questions of which 20 addressed the physical impact component and 9 assessed the psychological impact. A combined score can be generated, or both components can be reported separately. The psychological wellbeing assessment portion of the MSIS-29 was comprised of 9 questions in which subjects rate the impact of MS on their day-to-day life from 1=no impact to 5=extreme impact. The total Psychological Score was calculated using following formula: sum of score for 9 questions - 9/0.36. The total score range ranges from 0-100 where, lower total score indicates less psychologically-related impact while a higher total score indicates greater psychologically-related impact on a subject's functioning.
Severity of relapses (residual disability (EDSS) after relapses) | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses the 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), where higher scores indicate worse neurological function. Change was calculated by subtracting retreatment baseline (annual visit prior to the retreatment start date) value from EDSS scores at specified time points.
Frequency of serious adverse events | 2 year (96 week) period, with planned extension for 5 year (240 week) period
  Frequency of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bø, MD, Phd, Study Director — Haukeland University Hospital; Anne Kristine Lehmann, MD, PhD, Study Chair — Haukeland University Hospital; Astrid Kittang, MD, PhD, Study Chair — Haukeland University Hospital; Einar Kristoffersen, MD, PhD, Study Chair — Haukeland University Hospital; Øivind Torkildsen, MD, PhD, Study Chair — Haukeland University Hospital; Trygve Holmøy, MD, PhD, Principal Investigator — University Hospital, Akershus; Margitta Kampman, MD, PhD, Principal Investigator — Tromsø University Hospital; Kathrine K Liane, MD, Principal Investigator — St. Olavs Hospital; Joachim Burman, MD, PhD, Principal Investigator — Akademiska sjukhuset, Uppsala; Morten Blinkenberg, MD, PhD, Principal Investigator — Rigshospitalet, Denmark; Jan Lycke, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (8):
- Rigshospitalet, Copenhagen, Denmark
- VUmc, Amsterdam, Netherlands
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Oslo
  - University Hospital of North Norway, Tromsø
  - St. Olav's University Hospital, Trondheim
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within publication of the results.
Access Criteria: Data access requests will be reviewed by the RAM-MS steering committee. Requestors will be required to sign a data access agreement.

REFERENCES:
- See also: Study site (in Norwegian) — http://www.ram-ms.no

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT03477500/Prot_SAP_000.pdf